CLINICAL TRIAL: NCT06309563
Title: Study on the Metabolic Effects of a Diet Replaced With Essential Amino Acids and Carboxylic Acids (EAA-AC) in Patients With Severe Obesity
Brief Title: Metabolic Effects of a Diet Replaced With Essential Amino Acids
Acronym: AMINOB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31J301
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Obesity Morbid; Weight Loss
Keywords: Muscle mass during weight loss
MeSH Terms: conditions — Obesity, Morbid; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aminoacids (Active Comparator): Patients with obesity treated with essential aminoacids (EAA-AC)
  Interventions: Dietary Supplement: Aminoacid supplementation
- Control (Placebo Comparator): Patients with obesity treated with placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Aminoacid supplementation — Low-calorie and low-protein diet + with 4 sachets of EEA-AC supplement per day for 2 weeks
  Other Names: EAA-AC; Controls
  Arms: Aminoacids
Dietary Supplement: Placebo — Low-calorie and low-protein diet + placebo for 2 weeks
  Arms: Control

SUMMARY:
The effectiveness of low-protein diets supplemented with essential aminoacid (EAA) formulas in genetic disorders of amino acid (AA) catabolism, such as maple syrup urine disease (MSUD), is widely recognized (Blackburn PR et al. 2017). The main aim of the present study is to evaluate a difference in the effectiveness of a multidisciplinary rehabilitation program in patients with high degree of obesity with and without supplementation of this new formula of amino acids (essential + tricarboxylic acids - EAA-AC). For this reason, patients of both sexes, aged between 45 and 65, suffering from high-grade obesity will be recruited in Piancavallo. The enrolled patients divided, randomly, into two groups will be given: EAA-AC group a low-calorie and low-protein diet integrated with 4 sachets of EAA-AC supplement per day; the control group will follow a low-calorie and low-protein diet only with placebo. The parameters considered, after two weeks of treatment, will be: weight loss; the maintenance/recovery of muscle mass assessed through changes in body composition and functional tests (Hand grip, 6MWT or TUG) but also through the analysis of mitochondrial function in PBMC and circulating levels of mtDNA; the improvement of the glucose picture and the lipid profile.

1 month after discharge, patients will carry out an outpatient check-up to evaluate the maintenance of muscle mass using impedance testing.

ELIGIBILITY:
Inclusion Criteria:

- Obesity (BMI >35kg/m2)

Exclusion Criteria:

* Type 2 diabetes mellitus
* Renal failure
* Heart failure (New York Heart Association NYHA, class IV)
* Liver cirrhosis
* Neoplasms
* Muscular or non-autonomic pathologies
* Neurological-neurodegenerative pathologies
* Cognitive decline
* Non-menopausal women.
* Patients who have undergone bariatric surgery in the previous 12 months
* Patients on pharmacological treatment for weight loss in the last three weeks
* Patients using vitamin and amino acid supplements in the last three weeks
* Patients on hormone therapy (e.g. L-thyroxine, testosterone).

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle mass | At baseline and at 2 weeks after start of intervention
  Change in muscle mass during weight loss assessed through changes in body composition

SECONDARY OUTCOMES:
6 minute walking test (6MWT) | At baseline and at 2 weeks after start of intervention
  Change in distance covered in 6 minutes of walking during weight loss

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Site Piancavallo, Oggebbio, Verbania, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nisoli E, Falcone S, Tonello C, Cozzi V, Palomba L, Fiorani M, Pisconti A, Brunelli S, Cardile A, Francolini M, Cantoni O, Carruba MO, Moncada S, Clementi E. Mitochondrial biogenesis by NO yields functionally active mitochondria in mammals. Proc Natl Acad Sci U S A. 2004 Nov 23;101(47):16507-12. doi: 10.1073/pnas.0405432101. Epub 2004 Nov 15. PMID 15545607